CLINICAL TRIAL: NCT04694196
Title: Clinical Study to Locate Occlusal Plane According to Anatomical Landmark in Mandible
Brief Title: Use of Anatomical Landmark in Locate Occlusal Plane.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hama University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HU16-7-2020RemPro
Record Dates: First submitted 2020-12-16; First posted 2021-01-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Dentulous

STUDY DESIGN:
Intervention Model Description: No evidence of infection or trauma in oral Negative history of TMJ disorders
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Locate occlusal plane (Experimental): Use anatomical landmark to locate OP in dentulous subjects.
  Interventions: Device: Dentulous subjects

INTERVENTIONS:
Device: Dentulous subjects — Determine the occlusal plane using CN in anterior border of ramus

SUMMARY:
Occlusal plane "the average plane established by the incisal and occlusal surfaces of the teeth -The glossary of prosthodontic terms. Generally, it is not a plane but represents the planar mean of the curvature of these surfaces".

Correct orientation of the occlusal plane plays a vital role in achieving optimal aesthetics, occlusal balance and function of complete dentures. Faulty orientation of occlusal plane in fixed or removable prostheses will affect the interaction between tongue and buccinator muscle resulting in food collection in sulcus and cheek or tongue biting.

The occlusal plane is normally established anteriorly according to aesthetics of patient and posteriorly parallel to camper's plane.

In the mandibular arch there are few landmarks which could be used to orient the occlusal plane like the retromolar pad, commissure of the lips and lateral borders of the tongue.

Various landmark have been used to orient the occlusal plane in the maxillary arch e.g. parotid papilla, hamular notch- incisive papilla plane, ala-tragus line.

There is no single method seems entirely accurate to locate the occlusal plane in edentulous patients. Therefore ,Investigators need a stable anatomic landmark can be used as a guide to determine occlusal plane (OP).

Material and Methods:

Forty Dentulous patients will be selected. All subjects had natural maxillary and mandibular teeth. In addition all subjects exhibited Class I skeletal and dental relationships with no prosthetic dental replacement. Subjects with Claa II or Class III relationships,fractured or abraded edges of the teeth,ankyloglossia and orthodontic treatment were excluded from the study. The mandibular posterior occlusal plane was determined according to the level of coronoid notch{CN} (greatest concavity anterior border of the ramus) by measure the distance between the occlusal plane and CN.

DETAILED DESCRIPTION:
The plane of occlusion refers to an imaginary surface that theoretically touches incisal edges of the incisors and the tips of the occluding surfaces of the posterior teeth". A plane usually signifies a flat surface; however, it is not so where the occlusal plane is concerned. Two areas comprising of anterior and posterior teeth constitute the occlusal plane and must be considered individually. Anterior tooth position is governed by esthetics, phonetics and the required anterior guidance. On the contrary, functional needs predominantly determine the position of posterior teeth and this position is also affected by the incorporation of the anteroposterior and mediolateral curves. Optimal function, aesthetics and phonetics following prosthodontic rehabilitation is dependent on the establishment of physiologically accurate vertical dimensions of occlusion, palatal contours, positioning of the teeth and the level of occlusal plane.

The occlusal plane orientation is lost in patients with mutilated dentitions or those rendered edentulous and needs to be re-established for optimal function and comfort.

Different intra- and extra-oral landmarks used by clinicians to define the level of the occlusal plane include the upper lip, corners of mouth, lateral margins of tongue, Camper's plane and interpupillary line, the parotid papilla and the retromolar pad (RMP).

Any discrepancy in establishing the optimal level of occlusal plane causes adverse effects on periodontal tissues in dentate individuals and may result in vague symptoms such as headaches, migraines or stiffened shoulders and in edentulous patients, compromising the stability of the prosthesis, ultimately leading to alveolar bone resorption.

A combination of various landmark along with a judicious clinical judgment should be taken into account for the location of the occlusal plane in edentulous patients.

If the level of occlusal plane is too high, the tongue is unable to lie on the lingual cusps of the mandibular denture teeth and hence, fails to counter the movement of the denture. It may also result in food accretion in the labial and lingual sulci. In contrast, a low level of occlusal plane will promote tongue and cheek biting. Therefore, it is mandatory for the prosthodontist to re-establish the lost occlusal plane, both while dealing with multiple long span posterior restorations as well as in complete denture prosthodontics.

Material and Methods:

Forty dentulous patients. The mandibular posterior occlusal plane was determined on the level of coronoid notch (CN) on the anterior part of ramus. Then We will measure the occlusal plane in all forty a participants determined to the level of CN at the anterior border of ramus in mandible.

Inclusion :

* Stable systemic health, including absence of a history of cardiovascular disease
* No evidence of infection or trauma in oral region
* Negative history of TMJ disorders
* All subjects had natural maxillary and mandibular teeth.
* All subjects exhibited Class I skeletal and dental relationships with no prosthetic dental replacement.

Exclusion criteria:

Subjects with Claa II or Class III relationships,fractured or abraded edges of the teeth,ankyloglossia and orthodontic treatment The mandibular posterior occlusal plane was determined according to the level of coronoid notch{CN} (greatest concavity anterior border of the ramus) by measure the distance between the occlusal plane a with ages beyond the accepted age range

ELIGIBILITY:
Inclusion :

* Stable systemic health, including absence of a history of cardiovascular disease
* No evidence of infection or trauma in oral region
* Negative history of TMJ disorders
* All subjects had natural maxillary and mandibular All subjects exhibited Class I skeletal and dental relationships with no prosthetic dental replacement.

Exclusion Criteria:

Subjects with Claa II or Class III relationships,fractured or abraded edges of the teeth,ankyloglossia and orthodontic treatment were excluded from the study.

Ages: 21 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Occlusal plane marker in mandible | Through study completion .an average one week
  We will measure the occlusal plane in all forty a participants determined by a horizontal ruler to the level of Coronoid Notch(CN) at the anterior border of ramus in mandible.the measure will be in Millimetre(mm)above, under or at the level of Coronoid Notch(CN).
Aesthetic of complete denture in edentulous patients. | After 1 month
  After delivery the dentures to patients..we will examine the aesthetic effect to participants throughout examine acceptable response for the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Fadi Jnaid, Damascus, Rif-dimashq Governorate, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jain R, Shigli K. An in vivo study to correlate the relationship of the extraoral and intraoral anatomical landmarks with the occlusal plane in dentulous subjects. Indian J Dent Res. 2015 Mar-Apr;26(2):136-43. doi: 10.4103/0970-9290.159138. PMID 26096105
- [Background] Lundquist DO, Luther WW. Occlusal plane determination. J Prosthet Dent. 1970 May;23(5):489-98. doi: 10.1016/0022-3913(70)90198-8. No abstract available. PMID 4908801
- [Background] Kazanoglu A, Unger JW. Determining the occlusal plane with the Camper's plane indicator. J Prosthet Dent. 1992 Apr;67(4):499-501. doi: 10.1016/0022-3913(92)90080-t. PMID 1507133
- [Background] Al Quran FA, Hazza'a A, Al Nahass N. The position of the occlusal plane in natural and artificial dentitions as related to other craniofacial planes. J Prosthodont. 2010 Dec;19(8):601-5. doi: 10.1111/j.1532-849X.2010.00643.x. Epub 2010 Nov 11. PMID 21070428
- [Background] Nissan J, Barnea E, Zeltzer C, Cardash HS. Relationship between occlusal plane determinants and craniofacial structures. J Oral Rehabil. 2003 Jun;30(6):587-91. doi: 10.1046/j.1365-2842.2003.01044.x. PMID 12787455
- [Background] Tsay TP, Oyen OJ. A study of the suitability of two methods used for describing the occlusal plane. Proc Natl Sci Counc Repub China B. 1992 Jul;16(3):126-33. PMID 1296213
- [Background] Karkazis HC, Polyzois GL. A study of the occlusal plane orientation in complete denture construction. J Oral Rehabil. 1987 Jul;14(4):399-404. doi: 10.1111/j.1365-2842.1987.tb00735.x. PMID 3305842
- [Background] Raza M, Ayub N, Imran M, Nawaz K, Sami A. Occlusal Plane Evaluation In Dentate Patients For Complete Denture Prosthodontic Practice. J Ayub Med Coll Abbottabad. 2020 Jan-Mar;32(1):54-57. PMID 32468756
- [Background] Javid NS. A technique for determination of the occlusal plane. J Prosthet Dent. 1974 Mar;31(3):270-2. doi: 10.1016/0022-3913(74)90195-4. No abstract available. PMID 4521346